CLINICAL TRIAL: NCT02849483
Title: Effect of Ramosetron on Postoperative Restoration of Bowel Motility After Gynecological Laparoscopic Surgery
Brief Title: Effect of Ramosetron on Bowel Motility After Gynecological Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Mi Kyeong Kim, Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KHUH 2016-05-201
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; digestive signs and symptoms; vomiting; antiemetics; nausea; ramosetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Signs and Symptoms, Digestive; Vomiting; Nausea | interventions — ramosetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramosetron (Experimental): 2 ml of normal saline iv before induction, ramosetron 0.3 mg iv at the end of surgery, ramosetron 0.6 mg added to the iv PCA(Patient-Controlled Analgesia)
  Interventions: Drug: Ramosetron
- Control (Placebo Comparator): dexamethasone 10 mg iv before induction, 2 ml of normal saline iv at the end of surgery, 4 ml of normal saline added to the iv PCA
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ramosetron — Administer 2 ml of normal saline iv before induction. Inject ramosetron 0.3 mg iv at the end of surgery. Add ramosetron 0.6 mg to the iv PCA.
  Other Names: Nasea
  Arms: Ramosetron
Drug: Normal saline — Administer dexamethasone 10 mg iv before induction. Inject 2 ml of normal saline iv at the end of surgery. Add 4 ml of normal saline to the iv PCA.
  Arms: Control

SUMMARY:
Ramosetron is effective in preventing postoperative nausea and vomiting. Several studies reported that ramosetron is also effective treatment of irritable bowel syndrome. The investigators examine the effect of ramosetron on postoperative bowel motility.

DETAILED DESCRIPTION:
Ramosetron, a new potent and long-acting selective 5-HT3(5-hydroxytryptamine3) receptor anatagonist, is effective for preventing postoperative nausea and vomiting. Also several studies reported that ramosetron is effective treatment of diarrhea-predominant irritable bowel syndrome because it inhibits the accelerated colonic transit, abnormal colonic water transport, defecation abnormality, and the lowered colonic perceptual threshold by corticotrophin-releasing hormone, There is no study about the effect of ramosetron used for preventing postoperative nausea and vomiting on postoperative bowel motility. In this study, the investigators examine the effect of ramosetron on postoperative bowel motility.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 yrs of age
* ASA(American Society of Anesthesiologists) physical status class I or II
* Scheduled for gynecological laparoscopic surgery

Exclusion Criteria:

* Allergic to study drugs
* Antiemetics or steroids use within 24 hrs prior to surgery
* Dependence upon opioids
* Insulin dependent Diabetes Mellitus
* Cardiovascular or pulmonary disease
* Renal or hepatic insufficiency
* BMI>=35kg/m2
* History of motion sickness or PONV
* Cigarette smoker
* Conversion to open laparotomy from laparoscopic surgery
* Pregnants

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time from surgery to the passage of first flatus | Within 10 days after surgery

SECONDARY OUTCOMES:
Time to first defecation | Within 10 days after surgery
Incidence of postoperative ileus | Within 10 days after surgery

OTHER OUTCOMES:
Incidence and severity of postoperative nausea | 0-6 hours, 6-24 hours, and 24-48 hours after surgery
Incidence and severity of postoperative vomiting | 0-6 hours, 6-24 hours, and 24-48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mi Kyeong Kim, M.D., Ph.D., Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang HY, Kim Y, You AH, Kim YJ, Kim MK. A randomized controlled trial of the effect of ramosetron on postoperative restoration of bowel motility after gynecologic laparoscopic surgery. Int J Gynaecol Obstet. 2022 Jul;158(1):172-178. doi: 10.1002/ijgo.13969. Epub 2021 Oct 16. PMID 34614204